CLINICAL TRIAL: NCT06942962
Title: Assessment of Lymphocyte Subset Functions in Children Admitted to Assiut University Children Hospital With Acute Hepatitis A Infection
Brief Title: Immunity With Acute Hepatits A
Acronym: Hepatitis A
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Adel Attia Massod, Assistant lecturer, Assiut University
Other Study IDs: Lymphocyte subset functions
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis A; Hepatitis A Virus
Keywords: Immunity with hepatitis A in children; Lymphocyte subset function in hepatitis A
MeSH Terms: conditions — Hepatitis A; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis A Virus (HAV) is a public health concern in Egypt, especially among children. Historically highly endemic, recent studies suggest a changing epidemiology. While improved socioeconomic conditions have reduced its spread, HAV remains prevalent, with over 50% of Egyptians exposed by age 15. Infection is often asymptomatic or mild in children but can be more severe with age. Prevention relies on improved sanitation and hygiene, with vaccin and recov

DETAILED DESCRIPTION:
Introduction

Hepatitis A virus (HAV) infection remains a significant public health concern in Egypt, particularly among children. Egypt has historically been considered an area of high endemicity for HAV infection, with the highest prevalence occurring in early childhood. Recent studies, however, suggest a shifting epidemiological pattern. An estimated 8-10 million people suffer from viral hepatitis in Egypt, with HAV being one of the major causative agents.

The seroprevalence of HAV antibodies among Egyptian children has shown significant variability in recent years, reflecting changes in socioeconomic conditions and public health measures.

A study conducted in 2008 found that 61.4% of Egyptian children aged 2.5-18 years were seropositive for HAV antibodies. This study revealed a significant increase in HAV seroprevalence with higher age and lower social class. (WHO EMRO | Seroprevalence of Hepatitis A Virus, n.d.)Notably, among children under 6 years old, 72.7% from high social classes were seronegative for HAV antibodies, compared to only 19.0% from low social classes. These findings suggest that improvements in socioeconomic conditions may be altering the epidemiological landscape of HAV in Egypt.

More recent data indicate that HAV infection remains prevalent in Egypt, with 50% or more of the Egyptian population exposed to HAV by the age of 15. This high rate of early childhood exposure has important implications for public health strategies and vaccination policies.

Hepatitis A in children is often asymptomatic or presents with mild, non-specific symptoms. However, the severity of the disease tends to increase with age. In symptomatic cases, children may experience fever, fatigue, nausea, abdominal pain, and jaundice. While most cases resolve spontaneously without complications, severe manifestations such as fulminant hepatitis and liver failure have been reported in Egypt.

The risk of complications appears to be influenced by various factors, including age, nutritional status, and pre-existing liver conditions. In Egypt, where chronic liver diseases due to hepatitis B and C are prevalent, superinfection with HAV can lead to more severe outcomes.

Given the high prevalence of HAV in Egypt, prevention strategies are crucial. Improved sanitation and hygiene practices have contributed to reducing HAV transmission. However, vaccination remains the most effective preventive measure.

Currently, hepatitis A vaccination is not part of the standard immunization program in Egypt. The decision to implement universal vaccination should be based on cost-effectiveness analyses and the changing epidemiology of HAV in the country. Some experts recommend vaccination for high social class children at the preschool period without prior testing for HAV antibodies, while for middle social class children, vaccination after testing for HAV antibodies is suggested The immune response to HAV infection plays a crucial role in disease progression and resolution. In acute HAV infection, both innate and adaptive immune responses are activated. Natural Killer (NK) cells, part of the innate immune system, show a significant increase in the initial phase of acute hepatitis A, suggesting an important role in the first line of defense.

The adaptive immune response, particularly T cell-mediated immunity, is critical for viral clearance and long-term protection. Recent studies have highlighted the dominance of CD4+ T helper cell responses during acute resolving HAV infection.

CD4+ T cells produce multiple cytokines when viremia first declines and play a crucial role in the termination of HAV infection. In contrast, HAV-specific CD8+ T cells often fail to display effector functions until after viremia and hepatitis begin to subside.

Humoral immunity also plays a significant role in HAV infection. IgM anti-HAV antibodies appear within a few days of symptom onset and generally become undetectable within 4 months. Anti-HAV IgG antibodies, on the other hand, persist for life, providing long-term protection against reinfection.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-15 years
* Confirmed diagnosis of acute hepatitis A infection (positive anti-HAV IgM)
* Admitted to the hospital for management of acute hepatitis A
* Parental/guardian consent and child assent (where appropriate) obtained

Exclusion Criteria:

* Known pre-existing liver disease or chronic hepatitis
* Immunodeficiency disorders or current immunosuppressive therapy
* Coinfection with other hepatotropic viruses (HBV, HCV, HEV)
* Severe malnutrition
* Recent blood transfusion (within 3 months)

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-15 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between lymphocyte subset levels and development of hepatic encephalopathy or fulminant hepatic failure | One year

REFERENCES:
- [Background] Yigit M, Kalayci F. Vaccination status and hepatitis A immunity in children: insights from a large-scale study in Turkey. BMC Infect Dis. 2025 Jan 14;25(1):61. doi: 10.1186/s12879-025-10458-9. PMID 39810097
- [Background] Malik H, Malik H, Uderani M, Berhanu M, Soto CJ, Saleem F. Fulminant Hepatitis A and E Co-infection Leading to Acute Liver Failure: A Case Report. Cureus. 2023 Apr 25;15(4):e38101. doi: 10.7759/cureus.38101. eCollection 2023 Apr. PMID 37252544
- [Background] Gabrielli F, Alberti F, Russo C, Cursaro C, Seferi H, Margotti M, Andreone P. Treatment Options for Hepatitis A and E: A Non-Systematic Review. Viruses. 2023 Apr 28;15(5):1080. doi: 10.3390/v15051080. PMID 37243166
- [Background] Fouad HM, Reyad EM, El-Din AG. Acute hepatitis A is the chief etiology of acute hepatitis in Egyptian children: a single-center study. Eur J Clin Microbiol Infect Dis. 2018 Oct;37(10):1941-1947. doi: 10.1007/s10096-018-3329-0. Epub 2018 Jul 20. PMID 30030693
- [Background] El-Mokhtar MA, Elkhawaga AA, Ahmed MSH, El-Sabaa EMW, Mosa AA, Abdelmohsen AS, Moussa AM, Salama EH, Aboulfotuh S, Ashmawy AM, Seddik AI, Sayed IM, Ramadan HK. High Incidence of Acute Liver Failure among Patients in Egypt Coinfected with Hepatitis A and Hepatitis E Viruses. Microorganisms. 2023 Nov 30;11(12):2898. doi: 10.3390/microorganisms11122898. PMID 38138042
- [Background] Elbahrawy A, Ibrahim MK, Eliwa A, Alboraie M, Madian A, Aly HH. Current situation of viral hepatitis in Egypt. Microbiol Immunol. 2021 Sep;65(9):352-372. doi: 10.1111/1348-0421.12916. Epub 2021 Aug 21. PMID 33990999
- [Background] Doss W, Hermez J, Atta H, Jabbour J. Towards a hepatitis-free Egypt: is this achievable? (Editorial). East Mediterr Health J. 2018 Sep 6;24(7):609-610. doi: 10.26719/2018.24.7.609. PMID 30370918
- [Background] Abosheaishaa H, Abdelghany A, Abdelhalim O, Mohamed I, Morsi S, Youssef M, Salem A, Bahbah AA, Shady A, Naguib MS, Nassar M, El-Kassas M. The Egyptian journey from having the highest prevalence of hepatitis C virus to being the first to achieve "gold tier" in conquering the disease. Proc (Bayl Univ Med Cent). 2024 Jul 22;37(5):877-883. doi: 10.1080/08998280.2024.2379185. eCollection 2024. PMID 39165801
- See also: Related Info — https://www.emro.who.int/emhj-volume-14-2008/volume-14-issue-5/seroprevalence-of-hepatitis-a-virus-antibodies-among-a-sample-of-egyptian-children.html
- See also: Related Info — https://doi.org/10.4103/2667-3592.301462
- See also: Related Info — https://doi.org/10.7759/CUREUS.38101
- See also: Related Info — https://doi.org/10.1186/S12879-025-10458-9